CLINICAL TRIAL: NCT00211263
Title: Bipolar Disorder Center for Pennsylvanians (BDCP) Research Study
Brief Title: Bipolar Disorder Research Study for Ages 12 and Older
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kupfer, David J., M.D. (Individual)
Collaborators: Bristol-Myers Squibb (Industry); Abbott (Industry); GlaxoSmithKline (Industry); Pfizer (Industry); Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ME# 02-385; SAP# 4100010612
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2005-06

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

ARMS (2):
- Enhanced Clinical Intervention (Experimental)
  Interventions: Behavioral: Enhanced Clinical Intervention; Drug: mood stabilizer
- Clinical Intervention (Active Comparator)
  Interventions: Drug: mood stabilizer

INTERVENTIONS:
Behavioral: Enhanced Clinical Intervention
  Arms: Enhanced Clinical Intervention
Drug: mood stabilizer

SUMMARY:
The Bipolar Disorder Center for Pennsylvanians aims to reduce significant differences in treatment results among Pennsylvanians with bipolar disorder, especially among youth, the elderly, rural residents, and African Americans who are less likely to receive adequate treatment, less likely to remain in treatment once identified, and less likely to have positive results if they remain in treatment. Half of the subjects receive either Guideline Intervention (GI) or Enhanced Clinical Intervention (ECI). ECI is a combination of information and support, such as education about bipolar disorder, the medications used to treat it, information about sleep practices and habits that affect quality of sleep, review of symptoms, medication side effects, and coping with side effects. It is predicted that Enhanced Clinical Intervention will be more effective in reducing the differences in results between those most at risk compared to mid-life Caucasians. The treatment study occurs at three sites across Pennsylvania and has emphasized the recruitment of African Americans, youth (ages 12 through 18), and adults over age 65.

DETAILED DESCRIPTION:
Bipolar disorder is one of the world's most disabling conditions, robbing sufferers of years of healthy functioning. The presence of bipolar disorder is not limited to any nation, race, age, gender, or socioeconomic status, and has a lifetime prevalence of 1% across all populations. While there do not appear to be disparities in who is at risk for bipolar disorder, there are marked disparities in who is likely to be diagnosed and treated. The average person with bipolar disorder waits ten years before receiving the correct diagnosis (National Depression and Manic-Depression Association, 2000). Once a diagnosis of bipolar disorder is made, there are equally marked disparities in treatment outcome.

Also known as manic-depressive illness, bipolar disorder is a recurrent and chronic mental condition associated with substantial morbidity and mortality. The stigma associated with open recognition of this disorder decreases the likelihood of accurate diagnosis and treatment. Considering the impact of this disorder on the most vulnerable populations (youth, elderly, rural populations, and minorities), the challenge is to understand and reverse the current public health crisis. This crisis has created an enormous financial burden on the health, welfare, and disability systems. At the same time, it reduces the likelihood of economic and social productivity that can be achieved by potentially productive individuals.

The primary objective of the study is to test an intervention to reduce health disparities related to bipolar disorder, a vastly more destructive and difficult to treat condition than previously realized. The outcomes of interest include accurate and timely diagnosis, adequacy of prescribed treatment, retention in treatment, suicidality, and a range of treatment benefits including health-related quality of life, employment, treatment satisfaction, medication adherence, utilization of lower levels of intervention (e.g., outpatients versus partial or inpatient care), and reduction of substance use, medical morbidity and mortality. Particular attention has been paid to the collection of service utilization data to track key health care and social services. Costs for medical and psychiatric treatment, medications, inpatient, rehabilitation, and emergency room services are being ascertained for cost assessment, and patients' mood functioning is being tracked to assess the overall effectiveness of the interventions. The study is also using state-of-the-art assessments of phenotypic clinical variables to develop clinically meaningful predictors of treatment response across the age spectrum and across diverse racial groups.

To characterize more precisely the phenotypic complexity of this disorder, we have developed a spectrum model of psychiatric illness using a broader conceptualization of mood disorders and an integrated view of common comorbidities, anchored in the Mood and Anxiety Spectrum Assessments (Cassano et al. 1997; Cassano et al in press). This refined description of patient variability (or phenotypes) should lead to improved understanding of the variability in treatment outcomes among patients suffering from bipolar disorder and eventually to creating appropriate first-line treatments for patients who present with specific clinical phenotypes.

Careful consideration of biological phenotypes, as represented in population pharmacokinetics, turns a second line of attack on the problem of tailoring treatments to patients' specific needs. A key correlate of treatment response that has never been examined in bipolar disorder is consistent and adequate medication exposure. Essential to understanding variability in treatment response is being able to distinguish true non-responders from those who never received adequate exposure to drug. Consistency of drug exposure can be determined using a combination of electronic monitoring of drug-taking and population pharmacokinetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 12 years.
* Able to give basic informed consent.
* Meets DSM-IV Criteria for Bipolar I, Bipolar II (if in the investigator's judgment long term treatment with a mood stabilizer is indicated), Bipolar NOS, or Schizoaffective Bipolar subtype.
* Because many adolescents have shorter periods of mania or hypomania than those required by the DSM-IV (at least 4 days for hypomania and 7 days for mania) adolescents are included who have a current episode of MDD and a history of episodes mania/hypomania that lasted for at least 2 days.

Exclusion Criteria:

* Unwilling or unable to comply with study requirements (e.g., complete study forms, attend scheduled evaluations).
* Not competent to provide informed consent in the opinion of the investigator.
* Mental retardation (IQ less than 70). Subjects suspected of mental retardation (e.g., chronic academic failure, multiple developmental delays) are evaluated using the Verbal Subtest of the Wechsler Intelligence test.
* Presence of schizophrenia, schizoaffective pervasive developmental disorder, current substance or alcohol dependence, and organic mental disorder. Substance dependence in early remission is not an exclusion criterion.
* Unstable medical illness or other medical contraindication to treatment with mood stabilizers, antidepressants or antipsychotic medications.
* Women who are planning to become pregnant, pregnant or breast-feeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750
Dates: Start 2003-11; Study Completion 2007-02

PRIMARY OUTCOMES:
Key outcomes among all enrollments are ascertained every two months and continue throughout the 48-month period of the study. Outcomes include symptom and psychosocial factors, treatment adherence, disease severity, and resource utilization.

SECONDARY OUTCOMES:
Blood samples are drawn for pharmacotherapy exposure studies for each subject 11 times during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: David J Kupfer, MD, Principal Investigator — University of Pittsburgh Medical Center, Western Psychiatric Institute and Clinic
Locations (3):
- United States (3):
  - DuBois Regional Medical Center, DuBois, Pennsylvania
  - Thomas Jefferson University University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Fagiolini A, Frank E, Turkin S, Houck PR, Soreca I, Kupfer DJ. Metabolic syndrome in patients with bipolar disorder. J Clin Psychiatry. 2008 Apr;69(4):678-9. doi: 10.4088/jcp.v69n0423c. No abstract available. PMID 18507490
- See also: Click here for more information about this study: Bipolar Disorder Center for Pennsylvanians research study — http://www.wpic.pitt.edu/stanley/8thbipconf/Sample%20Abstract.doc